CLINICAL TRIAL: NCT01437540
Title: A Long-Term, Randomized, Study of the Safety and Tolerability of a Fixed-Dose Combination of Aclidinium Bromide/Formoterol Fumarate Compared With Formoterol Fumarate in Patients With Moderate to Severe, Stable Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Safety and Tolerability of Aclidinium Bromide/Formoterol Fumarate Compared With Formoterol Fumarate in Patients With Moderate to Severe Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LAC-MD-32
Record Dates: First submitted 2011-09-19; First posted 2011-09-21 (Estimated); Results first posted 2017-05-11 (Actual); Last update posted 2017-05-11 (Actual); Status verified 2017-03

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; Chronic Obstructive Pulmonary Disease; Chronic Bronchitis; Emphysema; Airflow Obstruction, Chronic; Chronic Airflow Obstruction; Chronic Obstructive Airway Disease; Chronic Obstructive Lung Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Bronchitis, Chronic; Emphysema | interventions — aclidinium bromide; Formoterol Fumarate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Inhaled aclidinium bromide 400 μg/formoterol fumarate 12 μg fixed dose combination (FDC), high dose twice per day
  Interventions: Drug: Aclidinium Bromide/Formoterol Fumarate
- 2 (Active Comparator): Inhaled formoterol fumarate 12 μg, twice per day
  Interventions: Drug: Formoterol Fumarate

INTERVENTIONS:
Drug: Aclidinium Bromide/Formoterol Fumarate — Inhaled aclidinium bromide 400 μg/formoterol fumarate 12 μg, high dose twice per day
  Arms: 1
Drug: Formoterol Fumarate — Inhaled formoterol fumarate 12 μg, twice per day
  Arms: 2

SUMMARY:
The purpose of this study is to assess the long-term safety and tolerability of inhaled aclidinium bromide/formoterol in patients with moderate to severe, stable chronic obstructive pulmonary disease (COPD).

ELIGIBILITY:
Inclusion Criteria:

* Current or former cigarette smokers with a cigarette smoking history of at least 10 pack-years
* A diagnosis of stable moderate to severe COPD and stable airway obstruction as defined by the Global Initiative for Chronic Obstructive Lung Disease guidelines and stable airway obstruction.

Exclusion Criteria:

* Patients who have been hospitalized for an acute COPD exacerbation within three months prior to Visit 1
* Any respiratory tract infection (including the upper respiratory tract) or COPD exacerbation in the six weeks before Visit 1.
* Patients with any clinically significant respiratory conditions other than COPD
* Clinical history that suggests that the patient has asthma as opposed to COPD
* Chronic use of oxygen therapy ≥ 15 hours/day
* Patients with clinically significant cardiovascular conditions
* Patients with uncontrolled infection that may place the patient at risk resulting from human immunodeficiency virus (HIV), active hepatitis and/or patients with diagnosed active tuberculosis
* Patients with a history of hypersensitivity reaction to inhaled anticholinergics,
* Patients with Stage II hypertension, defined as systolic pressure of 160 and above, and/or diastolic pressure of 100 and above
* Current diagnosis of cancer other than basal or squamous cell skin cancer

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 590 (Actual)
Dates: Start 2011-09-19 (Actual); Primary Completion 2013-03-31 (Actual); Study Completion 2013-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Esther Garcia, MD, Study Director — AstraZeneca
Locations (137):
- United States (137):
  - Forest Investigative Site 1162, Birmingham, Alabama
  - Forest Investigative Site 1493, Birmingham, Alabama
  - Forest Investigative Site 1620, Birmingham, Alabama
  - Forest Investigative Site 1127, Mobile, Alabama
  - Forest Investigative Site 1613, Chandler, Arizona
  - Forest Investigative Site 1623, Peoria, Arizona
  - Forest Investigative Site 1582, Phoenix, Arizona
  - Forest Investigative Site 1379, Phoenix, Arizona
  - Forest Investigative Site 1581, Phoenix, Arizona
  - Forest Investigative Site 1571, Phoenix, Arizona
  - Forest Investigative Site 1596, Fort Smith, Arkansas
  - Forest Investigative Site 1547, Encinitas, California
  - Forest Investigative Site 1088, Lakewood, California
  - Forest Investigative Site 1624, Los Angeles, California
  - Forest Investigative Site 1927, Los Angeles, California
  - Forest Investigative Site 1388, Paramount, California
  - Forest Investigative Site 1503, San Diego, California
  - Forest Investigative Site 1374, Torrance, California
  - Forest Investigative Site 1331, Vista, California
  - Forest Investigative Site 2039, Walnut Creek, California
  - Forest Investigative Site 1597, Boulder, Colorado
  - Forest Investigative Site 1137, Colorado Springs, Colorado
  - Forest Investigative Site 0892, Denver, Colorado
  - Forest Investigative Site 2037, Fort Collins, Colorado
  - Forest Investigative Site 1327, Wheat Ridge, Colorado
  - Forest Investigative Site 2045, Wheat Ridge, Colorado
  - Forest Investigative Site 1589, Norwalk, Connecticut
  - Forest Investigative Site 1598, Stamford, Connecticut
  - Forest Investigative Site 1154, Brandon, Florida
  - Forest Investigative Site 1944, Brandon, Florida
  - Forest Investigative Site 1152, Clearwater, Florida
  - Forest Investigative Site 1617, DeBary, Florida
  - Forest Investigative Site 1959, DeBary, Florida
  - Forest Investigative Site 1516, Edgewater, Florida
  - Forest Investigative Site 1403, Hollywood, Florida
  - Forest Investigative Site 1556, Orlando, Florida
  - Forest Investigative Site 1542, Ormond Beach, Florida
  - Forest Investigative Site 0974, Pensacola, Florida
  - Forest Investigative Site 2047, Tampa, Florida
  - Forest Investigative Site 1565, Venice, Florida
  - Forest Investigative Site 1851, Atlanta, Georgia
  - Forest Investigative Site 0980, Atlanta, Georgia
  - Forest Investigative Site 1567, Atlanta, Georgia
  - Forest Investigative Site 1607, Lawrenceville, Georgia
  - Forest Investigative Site 1409, O'Fallon, Illinois
  - Forest Investigative Site 2051, River Forest, Illinois
  - Forest Investigative Site 1604, Springfield, Illinois
  - Forest Investigative Site 1576, Evansville, Indiana
  - Forest Investigative Site 1549, Council Bluffs, Iowa
  - Forest Investigative Site 2033, Bowling Green, Kentucky
  - Forest Investigative Site 2085, Crescent Springs, Kentucky
  - Forest Investigative Site 1336, Louisville, Kentucky
  - Forest Investigative Site 2024, Lafayette, Louisiana
  - Forest Investigative Site 1430, New Orleans, Louisiana
  - Forest Investigative Site 1360, Sunset, Louisiana
  - Forest Investigative Site 1566, Auburn, Maine
  - Forest Investigative Site 1333, Baltimore, Maryland
  - Forest Investigative Site 1622, Columbia, Maryland
  - Forest Investigative Site 1590, Towson, Maryland
  - Forest Investigative Site 1570, Fall River, Massachusetts
  - Forest Investigative Site 1546, Haverhill, Massachusetts
  - Forest Investigative Site 1029, North Dartmouth, Massachusetts
  - Forest Investigative Site 1595, Worcestor, Massachusetts
  - Forest Investigative Site 1605, Traverse City, Michigan
  - Forest Investigative Site 1527, Fridley, Minnesota
  - Forest Investigative Site 1124, Minneapolis, Minnesota
  - Forest Investigative Site 1619, Plymouth, Minnesota
  - Forest Investigative Site 1587, Chesterfield, Missouri
  - Forest Investigative Site 1572, Jefferson City, Missouri
  - Forest Investigative Site 1399, St Louis, Missouri
  - Forest Investigative Site 1599, St Louis, Missouri
  - Forest Investigative Site 1831, Bozeman, Montana
  - Forest Investigative Site 1400, Missoula, Montana
  - Forest Investigative Site 1609, Bellevue, Nebraska
  - Forest Investigative Site 1616, Lincoln, Nebraska
  - Forest Investigative Site 1615, Omaha, Nebraska
  - Forest Investigative Site 1562, Las Vegas, Nevada
  - Forest Investigative Site 1610, Rochester, New Hampshire
  - Forest Investigative Site 1558, Brick, New Jersey
  - Forest Investigative Site 1559, Cherry Hill, New Jersey
  - Forest Investigative Site 1394, Ocean City, New Jersey
  - Forest Investigative Site 2084, Summit, New Jersey
  - Forest Investigative Site 0972, Brooklyn, New York
  - Forest Investigative Site 1163, New York, New York
  - Forest Investigative Site 1425, New York, New York
  - Forest Investigative Site 1554, Newburgh, New York
  - Forest Investigative Site 1563, Syracuse, New York
  - Forest Investigative Site 1557, Raleigh, North Carolina
  - Forest Investigative Site 1588, Shelby, North Carolina
  - Forest Investigative Site 1553, Wilmington, North Carolina
  - Forest Investigative Site 1550, Winston-Salem, North Carolina
  - Forest Investigative Site 1134, Canton, Ohio
  - Forest Investigative Site 1594, Cincinnati, Ohio
  - Forest Investigative Site 2028, Cincinnati, Ohio
  - Forest Investigative Site 1541, Marion, Ohio
  - Forest Investigative Site 1530, Toledo, Ohio
  - Forest Investigative Site 1393, Zanesville, Ohio
  - Forest Investigative Site 1612, Ashland, Oregon
  - Forest Investigative Site 1575, Corvallis, Oregon
  - Forest Investigative Site 1081, Eugene, Oregon
  - Forest Investigative Site 1580, Portland, Oregon
  - Forest Investigative Site 1552, Portland, Oregon
  - Forest Investigative Site 1574, Beaver, Pennsylvania
  - Forest Investigative Site 1577, Beaver, Pennsylvania
  - Forest Investigative Site 1126, Bethlehem, Pennsylvania
  - Forest Investigative Site 1423, Erie, Pennsylvania
  - Forest Investigative Site 1504, Hershey, Pennsylvania
  - Forest Investigative Site 1569, Pittsburgh, Pennsylvania
  - Forest Investigative Site 1548, Pittsburgh, Pennsylvania
  - Forest Investigative Site 1146, Pittsburgh, Pennsylvania
  - Forest Investigative Site 1560, Pittsburgh, Pennsylvania
  - Forest Investigative Site 1449, Tipton, Pennsylvania
  - Forest Investigative Site 1564, Uniontown, Pennsylvania
  - Forest Investigative Site 1144, Johnston, Rhode Island
  - Forest Investigative Site 2072, Charleston, South Carolina
  - Forest Investigative Site 1568, Easley, South Carolina
  - Forest Investigative Site 1506, Greenville, South Carolina
  - Forest Investigative Site 1601, Greer, South Carolina
  - Forest Investigative Site 0900, Spartanburg, South Carolina
  - Forest Investigative Site 1450, Union, South Carolina
  - Forest Investigative Site 1365, Rapid City, South Dakota
  - Forest Investigative Site 1440, Arlington, Texas
  - Forest Investigative Site 1954, Austin, Texas
  - Forest Investigative Site 1155, Dallas, Texas
  - Forest Investigative Site 1328, Dallas, Texas
  - Forest Investigative Site 1332, El Paso, Texas
  - Forest Investigative Site 2012, Fort Worth, Texas
  - Forest Investigative Site 1902, Killeen, Texas
  - Forest Investigative Site 1498, San Antonio, Texas
  - Forest Investigative Site 1614, San Antonio, Texas
  - Forest Investigative Site 1906, San Antonio, Texas
  - Forest Investigative Site 2004, San Antonio, Texas
  - Forest Investigative Site 1600, Magna, Utah
  - Forest Investigative Site 1480, Abingdon, Virginia
  - Forest Investigative Site 1579, Alexandria, Virginia
  - Forest Investigative Site 1142, Spokane, Washington
  - Forest Investigative Site 1573, Spokane, Washington

REFERENCES:
- [Derived] Donohue JF, Soong W, Wu X, Shrestha P, Lei A. Long-term safety of aclidinium bromide/formoterol fumarate fixed-dose combination: Results of a randomized 1-year trial in patients with COPD. Respir Med. 2016 Jul;116:41-8. doi: 10.1016/j.rmed.2016.05.007. Epub 2016 May 7. PMID 27296819
- See also: lac-md-32-synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=4061&filename=lac-md-32-synopsis.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 127 centers in the United States
  The first patient was screened in September 2011 and the last patient visit was in March 2013
Pre-assignment Details: The study consisted of a 2- to 3-week run-in period designed to assess the stability of patients' disease and establish each patient's baseline characteristics
  1063 patients were screened for eligibility; 473 were considered screen failures (main reason [406/473] inclusion/exclusion criteria not met)
Groups:
- Aclidinium/Formoterol 400 μg/12 μg: Aclidinium bromide/formoterol 400 μg/12 μg administered BID via dry-powder inhaler
- Formoterol 12 μg: Formoterol 12 μg administered BID via dry-powder inhaler
Period: Overall Study
Arm/Group | Aclidinium/Formoterol 400 μg/12 μg | Formoterol 12 μg
Started | 392 | 198
Completed | 265 | 133
Not Completed | 127 | 65
Not completed — Not listed below | 7 | 6
Not completed — COPD exacerbation | 13 | 3
Not completed — Lost to Follow-up | 3 | 5
Not completed — Lack of Efficacy | 23 | 11
Not completed — Protocol Violation | 24 | 12
Not completed — Adverse Event | 26 | 13
Not completed — Withdrawal by Subject | 31 | 15

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aclidinium/Formoterol 400 μg/12 μg | Formoterol 12 μg | Total
Number analyzed (Participants) | 392 | 198 | 590
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.9 (9.3) | 64.7 (9.4) | 64.2 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 176 | 89 | 265
  Male | 216 | 109 | 325

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients to Experience at Least One Treatment-emergent Adverse Event (TEAE)
Description: TEAEs were coded Version 16.0 of the Medical Dictionary for Regulatory Activities (MedDRA)
Time Frame: Up to study Week 56 ± 3 days
Population: Safety Population defined as all randomized patients who took at least one dose of double-blind investigational product
Measure: Number; unit: Percentage of participants
Arm/Group | Aclidinium/Formoterol 400 μg/12 μg | Formoterol 12 μg
Number analyzed (Participants) | 392 | 198
Percentage of participants | 71.4 | 65.7

2. Secondary Outcome: Percentage of Patients to Experience Any Potentially Clinically Significant (PCS) Post-baseline Change in Clinical Laboratory Values for Hematology, Chemistry or Urinalysis at the End of the Study
Description: <0.85 x lower limit of normal (LLN) or > 1.15 upper limit of normal (ULN) for hemoglobin, hematocrit, red blood cell, platelet, white blood cell, neutrophil and lymphocyte counts >1.15 × ULN for eosinophil, basophil and monocyte counts
  >1.15 x ULN for aspartate aminotransferase, alanine aminotransferase, alkaline phosphatase, gamma glutamyl transferase, total bilirubin, creatinine kinase, lactate dehydrogenase, blood urea nitrogen, creatinine, uric acid, total cholesterol, triglycerides <0.85 x LLN or >1.15 ULN for fasting glucose, calcium, phosphorus, total protein and albumin <0.95 x LLN or >1.05 x ULN for sodium, potassium and chloride
  Urinary blood, ketones or pH <0.85 x LLN or > 1.15 ULN
Time Frame: Up to study Week 52
Population: Patients with available non-potentially clinically significant baseline value and at least one post-baseline assessment
Measure: Number; unit: Percentage of participants
Arm/Group | Aclidinium/Formoterol 400 μg/12 μg | Formoterol 12 μg
Number analyzed (Participants) | 380 | 195
Percentage of participants | 63.9 | 62.1

3. Secondary Outcome: Percentage of Patients to Experience a Potentially Clinically Significant (PCS) Change in Pulse Rate, Systolic and Diastolic Blood Pressure
Description: Systolic BP ≥180 mmHg and increase ≥20 mmHg from baseline or ≤90 mmHg and decrease ≥20 mmHg from baseline; Diastolic BP ≥105 mmHg and increase ≥15 mmHg from baseline or ≤50 mmHg and decrease ≥15 mmHg from baseline; Pulse rate ≥ 110 bpm and increase ≥ 15% from baseline or ≤ 50 bpm and decrease ≥15% from baseline
Time Frame: Up to study Week 56 ± 3 days
Population: Patients with baseline and at least 1 post-baseline assessment of vital signs for each parameter
Measure: Number; unit: Percentage of patients
Arm/Group | Aclidinium/Formoterol 400 μg/12 μg | Formoterol 12 μg
Number analyzed (Participants) | 389 | 198
Percentage of patients
  Systolic BP ≥180 mmHg and increase ≥20 mmHg | 0.3 | 0.5
  Systolic BP ≤90 mmHg and decrease ≥20 mmHg | 1.5 | 1.0
  Diastolic BP ≥105 mmHg and increase ≥15 mmHg | 0 | 0.5
  Diastolic BP ≤50 mmHg and decrease ≥15 mmHg | 0.3 | 1.0
  Pulse rate ≥ 110 bpm and increase ≥ 15% | 0.8 | 0.5
  Pulse rate ≤ 50 bpm and decrease ≥15% | 0 | 0

4. Secondary Outcome: Percentage of Patients to Experience Potentially Clinically Significant Changes in ECG From Baseline
Description: Potentially clinically significant changes were defined as listed in the table below for QT interval, QTcB, QTcF, QRS interval, PR interval and heart rate (HR)
Time Frame: Up to study Week 56 ± 3 days
Population: Patients with baseline and at least 1 post-baseline assessment value for each parameter
Measure: Number; unit: Percentage of patients
Arm/Group | Aclidinium/Formoterol 400 μg/12 μg | Formoterol 12 μg
Number analyzed (Participants) | 392 | 198
Percentage of patients
  QT interval change from baseline >30 msec | 42.0 | 44.7
  QT interval >480 msec | 3.9 | 2.0
  QTcB change from baseline >30 msec | 31.1 | 30.3
  QTcB value >480 msec | 3.1 | 4.5
  QTcF change from baseline >30 msec | 21.5 | 22.7
  QTcF value >480 msec | 1.5 | 1.5
  QRS interval ≥100 msec and increase ≥25% from base | 2.0 | 1.0
  PR interval ≥200 msec and increase ≥25% from base | 2.8 | 1.0
  HR ≥110 bpm and decrease ≥15% from baseline | 2.6 | 1.0
  HR ≤50 bpm and decrease ≥15% from baseline | 4.6 | 4.0

ADVERSE EVENTS:
Time Frame: Up to study Week 56 ± 3 days
Arm/Group | Aclidinium/Formoterol 400 μg/12 μg | Formoterol 12 μg
Serious Adverse Events (participants affected / at risk) | 38/392 | 21/198
Other Adverse Events (participants affected / at risk) | 164/392 | 88/198
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aclidinium/Formoterol 400 μg/12 μg (N=392) | Formoterol 12 μg (N=198)
Pneumonia (Infections and infestations) | 4 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 1
Atrial fibrillation (Cardiac disorders) | 2 | 1
Death (General disorders) | 2 | 0
Non-cardiac chest pain (General disorders) | 2 | 0
Abscess intestinal (Infections and infestations) | 1 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Angina pectoris (Cardiac disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Atrial flutter (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 1
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0
Carotid artery disease (Nervous system disorders) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Completed suicide (Psychiatric disorders) | 1 | 0
Coronary artery occlusion (Cardiac disorders) | 1 | 0
Cystocele (Reproductive system and breast disorders) | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 1
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Hilar lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Lobar pneumonia (Infections and infestations) | 1 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Lung adenocarcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung carcinoma cell type unspecified stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Melaena (Gastrointestinal disorders) | 1 | 0
Mesenteric artery stenosis (Gastrointestinal disorders) | 1 | 0
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Peripheral vascular disorder (Vascular disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0
Rectocele (Reproductive system and breast disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Sarcoidosis (Immune system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Urinary retention postoperative (Injury, poisoning and procedural complications) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 1
Uterine prolapse (Reproductive system and breast disorders) | 1 | 0
VIIth nerve paralysis (Nervous system disorders) | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 1 | 0
Aortic stenosis (Vascular disorders) | 0 | 1
Brain mass (Nervous system disorders) | 0 | 1
Calculus ureteric (Renal and urinary disorders) | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 0 | 1
Chemical burn of skin (Injury, poisoning and procedural complications) | 0 | 1
Colonic stenosis (Gastrointestinal disorders) | 0 | 1
Convulsion (Nervous system disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Femoral hernia, obstructive (Gastrointestinal disorders) | 0 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Inguinal hernia, obstructive (Gastrointestinal disorders) | 0 | 1
Intestinal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Liver abscess (Infections and infestations) | 0 | 1
Mitral valve stenosis (Cardiac disorders) | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Vision blurred (Eye disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Aclidinium/Formoterol 400 μg/12 μg (N=392) | Formoterol 12 μg (N=198)
Nausea (Gastrointestinal disorders) | 7 | 11
Nasopharyngitis (Infections and infestations) | 25 | 9
Sinusitis (Infections and infestations) | 20 | 11
Upper respiratory tract infection (Infections and infestations) | 18 | 12
Urinary tract infection (Infections and infestations) | 26 | 11
Anxiety (Psychiatric disorders) | 23 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 10 | 10
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 106 | 57

LIMITATIONS AND CAVEATS:
The objective of the study is to assess the long-term safety and tolerability of inhaled aclidinium bromide/formoterol fixed-dose combination (FDC) Therefore there were were no primary and secondary efficacy assessments

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication of the results by the principal investigator (PI) will be subject to mutual agreement between the PI and sponsor